CLINICAL TRIAL: NCT00546390
Title: Protection of the Heart With Remote Ischemic Preconditioning During Heart Surgery: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Barry Finegan, MB, FFARC, FRCPC, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Protect
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Remote Ischemic Preconditioning; Myocardial Protection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ischemic Preconditioned Group (rIP) (Experimental): A 15-cm sterile blood pressure cuff was placed around the right thigh and connected to the inflating device, and the patient was draped obscuring the visibility of the cuff. Subsequently, the patient was randomly allocated (by opening of an envelope) to RIPC consisting of four 5-min cycles of lower limb ischemia-reperfusion induced by a tourniquet inflated to 300 mmHg
  Interventions: Device: Blood Pressure Cuff
- No Cuff (No Intervention): No rIP

INTERVENTIONS:
Device: Blood Pressure Cuff — The blood pressure cuff will be inflated for 5 minutes and then deflated for 5 minutes. This will be done 4 times in a row.
  Arms: Ischemic Preconditioned Group (rIP)

SUMMARY:
The purpose of this study is to compare a treatment called remote ischemic preconditioning (rIP) to no treatment. rIP is a simple treatment that is believed to help patients recover better after heart surgery. This treatment involves applying a large blood pressure cuff to one leg. The blood pressure cuffs will be inflated for 5 minutes and then deflated for 5 minutes. This will be done 4 times in a row.

DETAILED DESCRIPTION:
Purpose:

1. Determine, in a pilot study, if surrogate markers of rIP can be detected in patients presenting for cardiac surgery. Specifically measure the effect of rIP on the expression profile of HSP-70, iNOS, PKC-E, p38 MAPK, PI3K, and sarcolemmal KATP
2. Determine if rIP influences the expression of genes known to influence substrate preference and thereby myocardial metabolism in patients undergoing heart surgery. Specifically the expression of HIF-1a, PPAR-a and AMPK

Hypothesis:

We hypothesize that rIP provides myocardial protection in patients presenting for heart surgery and that this protection is defined by a distinct gene expression profile with regards to genes involved in rIP and myocardial metabolism.

Study Design:

This proposal is for a randomized blinded pilot study on the use of rIP in patients requiring heart surgery.

Study Population:

The study will include 100 male and female patients undergoing elective heart surgery with cardiopulmonary bypass (CPB).

Randomization:

Patients will be randomized 1:1 to receive either rIP or no treatment.

Blinding Procedures:

The patient will be blinded as well as those performing the experimental analysis.

Interventions:

Remote Ischemic Preconditioning

rIP will be induced immediately following induction of anesthesia. Four 5 minute cycles of lower unilateral limb ischemia and reperfusion induced tourniquet inflation to 300 mmHg will constitute the preconditioning stimulus.

Blood sample collection/analysis

1. Two cardiac biopsies (50 - 200 mg) will be collected pre-bypass and post- bypass and will be analyzed for gene and protein expression.
2. Blood samples (4 mL) will be drawn immediately before induction of anesthesia, and at the same times as cardiac tissue samples are harvested and analyzed for gene/protein expression as well as at 1, 24, 48 and 72 hours post surgery. Troponin I and NT-ProBNP will be measured at baseline, 1, 24, 48 and 72 hours after surgery and 3 mL of blood will be collected for these tests. A total of 43 mL of blood will be collected per patient.
3. rIP induced changes in leukocyte gene expression will be measured at the aforementioned time points.

Other

ECG assessment on post-operative day 1, 2, and 3.

National Institute of Health stroke scale assessment will be conducted at screening and post operatively prior to hospital discharge.

Each patient will receive a telephone follow-up call at 30 days post operatively to collect adverse events and mortality data.

Experimental Methods:

1. qRT-PCR will be used to measure gene expression.
2. Immunoblotting will be used to measure protein expression

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 through 80 years, inclusive
* Scheduled for heart surgery with CPB

Exclusion Criteria:

* Females of childbearing potential
* Emergency surgery
* Previous sternotomy
* Myocardial infarction within 48 hours prior to surgery
* Diabetes and/or BMI >35
* Need for Alpha2-agonists perioperatively
* Peripheral Vascular Disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Finegan, MB, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lucchinetti E, Bestmann L, Feng J, Freidank H, Clanachan AS, Finegan BA, Zaugg M. Remote ischemic preconditioning applied during isoflurane inhalation provides no benefit to the myocardium of patients undergoing on-pump coronary artery bypass graft surgery: lack of synergy or evidence of antagonism in cardioprotection? Anesthesiology. 2012 Feb;116(2):296-310. doi: 10.1097/ALN.0b013e318242349a. PMID 22222469
- See also: PubMed link — https://www.ncbi.nlm.nih.gov/pubmed/?term=Remote+Ischemic+Preconditioning+Applied+during++Isoflurane+Inhalation+Provides+No+Benefit+to+the++Myocardium+of+Patients+Undergoing+On-pump+Coronary++Artery+Bypass+Graft+Surgery

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 patients were withdrawn for logistical reasons
Groups:
- Placebo: No rIP - cuff placed but not used - actions by RA as if cuff inflated
Period: Overall Study
Arm/Group | Ischemic Preconditioned Group (rIP) | Placebo
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: No rIP as described for rIP group
- Total: Total of all reporting groups
Arm/Group | Ischemic Preconditioned Group (rIP) | Placebo | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 15 | 28
  >=65 years | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (7) | 62 (10) | 61 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 26 | 24 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Protection Against Ischemic Injury
Description: High-sensitivity cardiac troponin T release as measured by peak hscTnT values and area-under-the-curve.
Time Frame: 72 hours post operatively
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Placebo: No cuff inflation
Arm/Group | Ischemic Preconditioned Group (rIP) | Placebo
Number analyzed (Participants) | 27 | 28
pg/ml | 298 (266) | 231 (133)

2. Secondary Outcome: All-cause Death and Cardiovascular Long-term Outcome
Description: Death and re-hospitalization due to any cause including heart and renal failure and new atrial fibrillation
Time Frame: 6-month cardiovascular outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Ischemic Preconditioned Group (rIP) | Placebo
Number analyzed (Participants) | 27 | 28
Participants | 0 | 1

ADVERSE EVENTS:
Arm/Group | Ischemic Preconditioned Group (rIP) | No Cuff
All-Cause Mortality (participants affected / at risk) | 0/27 | 1/28
Serious Adverse Events (participants affected / at risk) | 3/27 | 3/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ischemic Preconditioned Group (rIP) (N=27) | No Cuff (N=28)
Heart Failure (Cardiac disorders) | 3 (3) | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
New Atrial Fib (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No